CLINICAL TRIAL: NCT00096694
Title: A Pilot Study Evaluating the Effect of the Levonorgestrel-Releasing Intrauterine Device on Genital HIV Shedding in HIV-1-Infected Women
Brief Title: Effect of an Intrauterine Contraceptive Device (IUD) in HIV Infected Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: A5205; 10187 (Registry Identifier: DAIDS ES); ACTG A5205
Record Dates: First submitted 2004-11-12; First posted 2004-11-15 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Intrauterine Device; IUD; Contraceptive; Levonorgestrel
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Device: Levonorgestrel-releasing intrauterine device (IUD)

SUMMARY:
Oral contraceptives (OCs) are not a good option for some HIV infected women because of the potential for drug interactions between OCs and anti-HIV drugs; additionally, OCs may increase the risk of transmitting HIV to sexual partners. Levonorgestrel is commonly prescribed as part of a combination OC. An intrauterine device (IUD) is a device inserted in a woman's uterus to prevent pregnancy. The purpose of this study is to determine the effect of a levonorgestrel-releasing IUD on the amount of HIV present in an HIV infected woman's cervix after 4 weeks of IUD use.

Study hypothesis: There will be no increase in genital tract HIV RNA and DNA after placement of the levonorgestrel IUD.

DETAILED DESCRIPTION:
HIV infected women face the challenges of preventing both pregnancy and HIV transmission to their sexual partners. However, OCs may interact with antiretroviral therapy (ART), and data suggest that higher doses of OCs may increase cervical shedding of HIV-1, which may increase an HIV infected woman's infectiousness to her sexual partners. A physical barrier contraceptive would be useful to HIV infected women to circumvent the problems associated with concurrent use of OCs and ART. The levonorgestrel IUD has proved highly effective in preventing unwanted pregnancies in HIV uninfected women since its introduction in the United States in 1999. This study will evaluate the effect of the levonorgestrel IUD on HIV viral load in an HIV infected woman's cervix after 4 weeks of IUD use.

This study will last approximately 48 weeks; there will be 4 study visits. At screening, participants will undergo medical and medication history assessment; a complete physical exam; a pelvic exam, including genital tract sample collection; blood collection; sexually transmitted disease (STD) testing; and a Pap smear, if needed. The levonorgestrel IUD will be inserted into the participant's uterus at study entry. At study entry and at Weeks 4, 16, and 48, participants will undergo a targeted physical exam; a pelvic exam, including genital tract sample collection; and blood collection. Participants will be given a menstrual diary at the start of the study and at each study visit and will be asked to document all menstrual cycles they have for the duration of the study.

To be eligible for this study, participants may not have had ART within 90 days prior to study entry. However, after the Week 4 study visit, participants may reinitiate (if they were on ART more than 90 days prior to study entry) or initiate (if they are ART naive) ART, if deemed necessary to do so by their physicians.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* Willing and able to delay initiation or reinitiation of antiretroviral therapy until after Week 4 study visit
* Unlikely to develop a clinical indication to start antiretroviral therapy within 4 weeks of study entry
* CD4 count of 200 cells/mm3 or more
* Viral load of 10,000 copies/ml or more within 90 days prior to study entry
* Endocervical viral load of 2,500 copies/ml or more within 90 days prior to study entry
* History of prior pregnancy lasting at least 20 weeks
* Willing to continue any current use of hormonal contraceptives, except medroxyprogesterone acetate, until after Week 4 study visit
* Start of last menstrual period within 7 days prior to study entry

Exclusion Criteria:

* Antiretroviral medications within 90 days prior to study entry
* AIDS diagnosis, including CD4 count of less than 200 cells/mm3
* Cervicitis, bacterial vaginosis, trichomoniasis, or symptomatic vaginal candidiasis within 90 days prior to study entry. Participants with any of these infections within 90 days prior to study entry are not excluded if they have received appropriate treatment and have documented resolution of the infection.
* Acute or history of pelvic inflammatory disease, chlamydia, or gonorrhea in the year prior to study entry
* Abnormal Pap smear requiring treatment in the year prior to study entry
* History of ectopic pregnancy or a condition that would predispose the participant to ectopic pregnancy
* Known uterine anomaly, including fibroids
* Known or suspected breast cancer
* Acute liver disease or liver tumor
* Have previously inserted IUD that has not been removed
* Fungal infection in the genitals
* Genital bleeding of unknown cause
* Endometritis or infected abortion within 90 days of study entry
* Known allergy or hypersensitivity to any component of the IUD used in this study
* Current drug or alcohol abuse that, in the opinion of the investigator, may interfere with the study
* Serious infection or other serious medical illness that is potentially life threatening and requires systemic therapy or hospitalization within 14 days of study entry
* Use of etonogestrel and ethinyl estradiol vaginal ring (NuvaRing) within 30 days prior to study entry
* Medroxyprogesterone acetate within 90 days prior to study entry
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41
Dates: Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Sign and magnitude of difference in endocervical HIV viral load from baseline to Week 4 post-IUD insertion
incidence of discontinuation of IUD use in the year following insertion

CONTACTS AND LOCATIONS:
Overall Officials: E. Milu Kojic, MD, Study Chair — Department of Immunology/Infectious Disease, The Miriam Hospital
Locations (9):
- United States (8):
  - UCLA CARE Center CRS, Los Angeles, California
  - IHV Baltimore Treatment CRS, Baltimore, Maryland
  - SSTAR, Family Healthcare Ctr., Fall River, Massachusetts
  - Washington U CRS, St Louis, Missouri
  - Beth Israel Med. Ctr., ACTU, New York, New York
  - Duke Univ. Med. Ctr. Adult CRS, Durham, North Carolina
  - Rhode Island Hosp., Providence, Rhode Island
  - The Miriam Hosp. ACTG CRS, Providence, Rhode Island
- Puerto Rico-AIDS CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] Bird ST, Harvey SM, Maher JE, Beckman LJ. Acceptability of an existing, female-controlled contraceptive method that could potentially protect against HIV: a comparison of diaphragm users and other method users. Womens Health Issues. 2004 May-Jun;14(3):85-93. doi: 10.1016/j.whi.2004.03.003. PMID 15193636
- [Background] Richardson BA, Morrison CS, Sekadde-Kigondu C, Sinei SK, Overbaugh J, Panteleeff DD, Weiner DH, Kreiss JK. Effect of intrauterine device use on cervical shedding of HIV-1 DNA. AIDS. 1999 Oct 22;13(15):2091-7. doi: 10.1097/00002030-199910220-00012. PMID 10546862
- [Background] Stuart GS, Castano PM. Sexually transmitted infections and contraceptives: selective issues. Obstet Gynecol Clin North Am. 2003 Dec;30(4):795-808. doi: 10.1016/s0889-8545(03)00074-3. PMID 14719851
- [Background] Wang CC, McClelland RS, Overbaugh J, Reilly M, Panteleeff DD, Mandaliya K, Chohan B, Lavreys L, Ndinya-Achola J, Kreiss JK. The effect of hormonal contraception on genital tract shedding of HIV-1. AIDS. 2004 Jan 23;18(2):205-9. doi: 10.1097/00002030-200401230-00009. PMID 15075537